CLINICAL TRIAL: NCT01850875
Title: Localized and Generalized Musculoskeletal Pain: Psychobiological Mechanisms and Implications for Treatment (LOGIN) - Subgroups Characterized by Psychological Trauma, Mental Comorbidity, and Psychobiological Patterns and Their Specialized Treatment - Eye Movement Desensitization and Reprocessing (EMDR) in Non-specific Chronic Back Pain
Brief Title: Eye Movement Desensitization and Reprocessing (EMDR) in Non-specific Chronic Back Pain
Acronym: LOGIN - EMDR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Heidelberg (Other)
Responsible Party: Principal Investigator, Prof. Dr. Wolfgang Eich, Prof. Dr., University Hospital Heidelberg
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 01EC1010A
Record Dates: First submitted 2013-04-23; First posted 2013-05-10 (Estimated); Last update posted 2016-05-16 (Estimated); Status verified 2016-05

CONDITIONS: Non-specific Chronic Back Pain
Keywords: Eye-Movement-Desensitization and Reprocessing; EMDR; Chronic back pain; CBP; treatment
MeSH Terms: interventions — Eye Movement Desensitization Reprocessing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Eye-Movement-Desensitization-Reprocessing (Experimental): Eye-Movement-Desensitization-Reprocessing
  Interventions: Behavioral: Eye-Movement-Desensitization-Reprocessing
- Treatment as usual (control group) (No Intervention): treatment as usual

INTERVENTIONS:
Behavioral: Eye-Movement-Desensitization-Reprocessing
  Arms: Eye-Movement-Desensitization-Reprocessing

SUMMARY:
The study explores the feasibility of Eye-Movement-Desensitization and Reprocessing (EMDR) in non-specific chronic back pain.

DETAILED DESCRIPTION:
The study explores the feasibility of Eye-Movement-Desensitization and Reprocessing (EMDR) in non-specific chronic back pain in a randomized controlled trial (RCT) with 6 months follow-up. The treatment consists of 12-sessions EMDR a 60 minutes using eye-movements for bilateral stimulation in addition to treatment as usual (TAU) that is compared to TAU alone.

ELIGIBILITY:
Inclusion Criteria:

* >= 18 years
* non-specific chronic low back pain >= 45 days/3 months
* high emotional distress caused by psychological trauma
* German language skills

Exclusion Criteria:

* specific causes of chronic back pain
* application for retirement pension pending
* ongoing psychotherapy
* severe physical or psychiatric comorbidity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-05; Primary Completion 2014-11 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change in pain intensity | Change from Baseline Pain intensity at average 6 months
  Numerical rating scale 0-10

OTHER OUTCOMES:
functional and structural changes in fMRI | Change from Baseline fMRI at average 6 months
Change in the pain experience scale - Pain affect | Change from Baseline pain experience scale levels at average 6 months
  Geisser et al., 1996
Change in the Hannover functional ability questionnaire (FFbH) - disability | Change from Baseline disabilty levels at average 6 months
  Kohlmann et al., 1996
Change in Quantitative sensory testing (QST)profiles | Change from Baseline QST profile at average 6 months
  According to the protocol by Rolke et al. (2006), developed within the Germany Research Network on Neuropathic Pain (DFNS)
Change in Conditioned Pain Modulation | Change from Baseline conditioned pain modulation activity at average 6 months
  difference in pressure pain threshold before and after oscillating heat (2 min.)
Change in Plasma endocannabinoids and lipids | Change from Baseline endocannabinoids and lipids at average 6 months
  Plasma levels: AEA (ng/ml), 2-AG (ng/ml), AA (ng/ml), PEA (ng/ml), OEA (ng/ml), AEA (pmol/g), 2-AG (pmol/g), AA (nmol/g), PEA (pmol/g), OEA (pmol/g),
Change in plasma nerve growth factor levels | Change from Baseline NGF levels at average 6 months
  Plasma levels in (pg/ml)
Change in pain drawing/ the spatial extent of the pain | Change from Baseline Pain extent at average 6 months
Change in West Haven-Yale multidimensional pain inventory scores | Change from Baseline West Haven-Yale multidimensional pain inventory scores at average 6 months
  Flor et al., 1990
Change in chronic pain grade | Change from Baseline chronic pain grade at average 6 months
  von Korff er al., 1992
Change in Resilience Scale (RS-11) scores | Change from Baseline resilience scores at average 6 months
  Schumacher et al., 2004
Change in Hospital Anxiety and Depression Scale scores | Change from Baseline anxiety and depression levels at average 6 months
  Zigmond & Snaith, 1983
Change in Health Survey scores | Change from baseline quality of life level at average 6 months
  SF-12
Change in somatization scores | Change from Baseline somatization scores at average 6 months
  SCL-90R
Change in medication intake | Change from Baseline medication intake at average 6 months
Change in dissociation scores | Change from Baseline dissociation at average 6 months
  DES/FDS-20
Change in Post Traumatic Diagnostic Scale | Change from Baseline post traumatic diagnostic scale levels at average 6 months
Patient global impression of change | after on average 6 months of treatment
Recruitment potential | 6 months
  % of patients eligible for inclusion that give written informed consent
Retention rate | over average 6 months of treatment
  % of patients that finish treatment, including pre- and post-evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Eich, Prof. Dr., Principal Investigator — University Hospital Heidelberg
Locations (1):
- University Hospital Heidelberg, Heidelberg, Baden-Wurttemberg, Germany

REFERENCES:
- [Derived] Gerhardt A, Leisner S, Hartmann M, Janke S, Seidler GH, Eich W, Tesarz J. Eye Movement Desensitization and Reprocessing vs. Treatment-as-Usual for Non-Specific Chronic Back Pain Patients with Psychological Trauma: A Randomized Controlled Pilot Study. Front Psychiatry. 2016 Dec 20;7:201. doi: 10.3389/fpsyt.2016.00201. eCollection 2016. PMID 28066274
- [Derived] Tesarz J, Gerhardt A, Leisner S, Janke S, Hartmann M, Seidler GH, Eich W. Effects of eye movement desensitization and reprocessing (EMDR) on non-specific chronic back pain: a randomized controlled trial with additional exploration of the underlying mechanisms. BMC Musculoskelet Disord. 2013 Aug 30;14:256. doi: 10.1186/1471-2474-14-256. PMID 23987561
- See also: Consortium LOGIN — http://www.login-verbund.de/index.php?id=2&L=1